CLINICAL TRIAL: NCT00228540
Title: An 8 Week, Open-Label Study to Characterize the Response to Modafinil (85 mg Film Coated Tablet) Treatment at Dosages Up to 425 mg/Day in Children and Adolescents With Attention Deficit/Hyperactivity Disorder (ADHD) (With an Open Ended Extension Period)
Brief Title: Study to Assess Satisfaction With Modafinil Treatment in Children and Adolescents With ADHD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cephalon (Industry)
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: C1538/3044/AD/US
Record Dates: First submitted 2005-09-27; First posted 2005-09-29 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-05

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Modafinil

INTERVENTIONS:
Drug: Modafinil

SUMMARY:
An 8-week, Open-Label Study to Characterize the Response to Modafinil (85mg Film-Coated Tablet) Treatment at Dosages up to 425mg/Day in Children and Adolescents with Attention-Deficit/Hyperactivity Disorder (ADHD) (With an Open-Ended Extension Period)

ELIGIBILITY:
Inclusion Criteria:

Patients are included in the study if all of the following criteria are met:

* Written informed consent/assent is obtained.
* The patient is a boy or girl 6 through 17 years of age (inclusive) at the screening visit, and both the patient and parent/legal guardian are English-speaking.
* The patient has a previous diagnosis of ADHD and is currently receiving medication for the treatment of ADHD.
* The patient, or the patient's parent/legal guardian, is dissatified (VAS score <50) with current ADHD medication (medication and reason for dissatisfaction documented).
* The patient is in good health as determined by a medical or psychiatric history, screening physical examination, and clinical laboratory evaluations.
* Girls who are postmenarche or sexually active, must have a negative urine pregnancy test prior to the baseline visit, must be using a medically acceptable method of birth control, and must agree to continue use of this method for the duration of the study (and for 30 days after participation in the study). Acceptable methods of birth control include the following: barrier method with spermicide; steroidal contraceptive (eg, oral, transdermal, implant, or injected) in conjunction with a barrier method; intrauterine device (IUD); and abstinence.
* The patient's parent/legal guardian must be willing and able to comply with study procedures and restrictions.

Exclusion Criteria:

Patients are excluded from participating in this study if 1 or more of the following criteria are met:

* The patient has any current psychiatric comorbidity, including but not limited to depression or other mood disorder, or pervasive mental disorder, that requires pharmacotherapy.
* The patient is satisfied with current ADHD medication and has no side effects.
* The patient is using other prescription medications for ADHD with psychoactive properties (eg, amphetamine, dextroamphetamine, methylphenidate, pemoline, atomoxetine) after the baseline visit.
* The patient has used monoamine oxidase (MAO) inhibitors within 1 week before the baseline visit.
* The patient has used an investigational drug within 1 month before the screening visit.
* The patient has a known clinically significant drug sensitivity to modafinil or any of its inactive ingredients.
* The patient is pregnant or lactating. (Any patients becoming pregnant during the study will be withdrawn from study).

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 2005-09; Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (39):
- United States (39):
  - Melmed Center, Scottsdale, Arizona
  - UCI Child Development Center, Irvine, California
  - Pharmacology Research Institut, Northridge, California
  - Pacific Sleep Medicine Service, San Diego, California
  - Sarkis Clinical Trials, Gainesville, Florida
  - Clinical Neuroscience Solution, Jacksonville, Florida
  - Clinical Neurosciences, Orlando, Florida
  - Laszlo J. Mate, MD, PA, West Palm Beach, Florida
  - Northwest Behavioral Research, Marietta, Georgia
  - Pediatrics and Adolescent, Woodstock, Georgia
  - Loyola University Medical Center Department of Psychiatry, Maywood, Illinois
  - HALP Clinic and ADHD Research, Northbrook, Illinois
  - Cientifica, Inc., Wichita, Kansas
  - Michael J. Rieser, MD, Lexington, Kentucky
  - Pedia Research, LLC, Owensboro, Kentucky
  - Louisiana Research Associates, New Orleans, Louisiana
  - Psycopharmacology Research - LSU Health Science Center, Shreveport, Louisiana
  - Massachusetts General Hospital, Cambridge, Massachusetts
  - Odyssey Research, Dearborn, Michigan
  - Hurley Medical Center, Flint, Michigan
  - ProMed HealthCare, Kalamazoo, Michigan
  - Regions Hospital, Saint Paul, Minnesota
  - Odyssey Research, McCook, Nebraska
  - University of Nebraska, Omaha, Nebraska
  - Bancroft Clinical Research, Cherry Hill, New Jersey
  - Hunterdon Pediatric Associates, Flemington, New Jersey
  - Odyssey Research, Bismarck, North Dakota
  - Prairie at Saint John's, Fargo, North Dakota
  - Odyssey Research, Minot, North Dakota
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - OCCI, Inc Salem, Salem, Oregon
  - Medical University of SC, Charleston, South Carolina
  - UT Medical Group, Memphis, Tennessee
  - Clinical Neuroscience Solution, Memphis, Tennessee
  - Claghorn-Lesem Research, Bellaire, Texas
  - The Clinical Study Ceneter, Burlington, Vermont
  - Dominion Clinical Research, Midlothian, Virginia
  - Advanced Pediatrics, Vienna, Virginia
  - Eastside Therapeutic Resource, Kirkland, Washington